CLINICAL TRIAL: NCT04757688
Title: RAD 1901: Noninvasive Cardiac Radioablation for Ventricular Tachycardia Refractory to Medication and Catheter Ablation
Brief Title: Noninvasive Cardiac Radioablation for Ventricular Tachycardia Refractory to Medication and Catheter Ablation
Acronym: RAD 1901
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with accrual
Sponsor: John Stahl (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, John Stahl, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006881
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Ventricular Tachycardia
Keywords: Cardiac radioablation; Cardiac SBRT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cardiac radioablation (CRA) (Experimental): CRA delivered via linear accelerator (stereotactic body radiotherapy) to the suspected arrhythmogenic substrate to a dose of 25 Gy in 1 fraction.
  Interventions: Radiation: Cardiac radioablation (CRA)

INTERVENTIONS:
Radiation: Cardiac radioablation (CRA) — CRA to 25 Gy in 1 fraction

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of cardiac radioablation (CRA) as a means of noninvasive treatment of ventricular tachycardia (VT) refractory to both medication and catheter ablation.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a regular, rapid (faster than 100 beats per minute) abnormal heart rhythm resulting from aberrant electrical conduction in the ventricles of the heart. Coronary heart disease is responsible for the majority of VT cases. Defibrillation and antitachycardia pacing, effective means of terminating a life-threatening acute episode of VT, can be delivered via implantable cardioverter-defibrillator (ICD). ICDs are able to both monitor the heart rhythm continuously and deliver therapy in response to tachycardia that meets pre-programmed detection criteria. For patients with VT refractory to medical management requiring multiple ICD shocks, electrophysiologic mapping may be utilized to localize the arrhythmogenic focus, which can be subsequently ablated with cardiac catheter radiofrequency ablation. The goal of catheter ablation is to identify (through electroanatomical mapping) and then eliminate the channels of surviving myocardium within the substrate. Many patients experience continued episodes of VT refractory to both medication and multiple catheter ablation attempts. ICD shocks are associated with substantially increased risk of hospitalization, quality of life impairment, and death.

Stereotactic body radiotherapy (SBRT) is a technique used most commonly as a cancer treatment, whereby a precise, high dose of radiation is delivered to a target. For patients with VT refractory to medication and catheter ablation, noninvasive targeting of the arrhythmogenic substrate with SBRT (in this case termed cardiac radioablation, CRA) is an emerging technique demonstrating favorable efficacy.

Using a protocol similar to that utilized by the phase I/II ENCORE-VT trial (NCT02919618), this study aims to replicate previously reported favorable results in a multi-institutional setting. Accrued patients will receive CRA to 25 Gy in a single fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old.
* Patients must have documented sustained monomorphic VT by 12-lead ECG or intracardiac ICD interrogation.

  * Minimum VT burden: 4 or more documented VT episodes (including sustained VT, ICD anti-tachycardia pacing [ATP], or ICD shock) in the 5 months preceding enrollment on this trial. Patients must have at least two episodes of electrocardiographically documented symptomatic, recurrent, sustained monomorphic VT in the 3 months prior to enrollment
  * *ATP and appropriate ICD shock are acceptable surrogates for VT-associated symptoms
* Patients must have an ICD.
* Patients must have ischemic or non-ischemic cardiomyopathy previously diagnosed with LVEF ≤ 35%.
* Patients must have received at least one antiarrhythmic medication (i.e. amiodarone, sotalol, mexiletine) without control of symptoms or with poor toleration. AND Patients must have undergone at least one catheter-ablation procedure (or have a contraindication to catheter-ablation) or have VT arising from an inaccessible location.

  * Contra-indications to endocardial catheter ablation procedure include dual aortic and mitral mechanical valves, active left ventricular thrombus, and anesthesia intolerance.
  * Contra-indications to epicardial catheter ablation include prior cardiac surgery or anesthesia intolerance.
  * Patients with ischemic cardiomyopathy should have failed at least one endocardial ablation performed at an academic center.
  * Patients with non-ischemic cardiomyopathy should have failed both epicardial and endocardial ablations, unless epicardial mapping/ablation is not feasible.
* Ability to understand and willingness to sign an IRB approved informed consent document (legally authorized representatives are not permissible).
* An independent EP cardiologist must confirm that each study participant has met the study entrance criteria, has failed conventional therapies, and has frequent recurrent VT episodes that warrant further rhythm management.

Exclusion Criteria:

* Patients who have received any prior radiotherapy to the internal organs of the thorax or upper abdomen (with treatment field extending superior to L1 vertebral body) at any time in the past are excluded.
* Patients found to have multiple scars on electrocardiographic imaging where the source of reentrant focus is unclear despite positron emission tomography (PET)/magnetic resonance imaging (MRI) are excluded.
* Patients who have congestive heart failure on inotropes (NYHA class 4B) or left-ventricular assist device are excluded.
* Patients felt to be unlikely to live 12 months in the absence of VT are excluded.
* Patients with polymorphic VT or ventricular fibrillation, >3 distinct clinical VT morphologies on ICD interrogation, or >5 induced VT morphologies during noninvasive testing are excluded.
* Patients with multiple, spatially separate target substrates (targets with presumed inclusion of nonadjacent ventricular segments) deemed unsafe to treat with CRA by the treating physician will be excluded.
* Patients with incessant VT that is hemodynamically unstable are excluded.
* Patients in VT storm are excluded.
* Patients must not be pregnant and must have a negative pregnancy test within 14 days of study entry if they are females of childbearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in ICD treatments for VT (≥ 50 percent) | 6 months
  Number of subjects with ≥ 50 percent reduction in number of ICD treatments for VT (shocks or anti-tachycardia pacing, ATP) comparing 5 month period before CRA to 6 months after CRA (excluding 1 month blanking period post CRA).

SECONDARY OUTCOMES:
Severe adverse event rate ≤ 20 percent | 3 months
  Demonstration of a ≤ 20 percent rate of severe adverse events within 90 days of CRA.
Reduction in ICD treatments for VT (≥ 95 percent) | 6 months
  Number of subjects with ≥ 95 percent reduction in number of ICD treatments (shocks or ATP) for VT comparing 5 month period before CRA to 6 months after CRA (excluding 1 month blanking period post CRA).
Elimination of ICD shocks | 5 years
  Number of subjects with elimination of ICD shocks.

CONTACTS AND LOCATIONS:
Overall Officials: John Stahl, MD, Principal Investigator — University of Alabama at Birmingham (UAB); Cliff Robinson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Alabama at Birmingham (UAB) Department of Radiation Oncology, Birmingham, Alabama, United States